CLINICAL TRIAL: NCT03180567
Title: Pharmacogentic Screening of Coumarine Based Oral Anticoagulant Using Next Generation Seguencer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Prof Amr gawaly
Record Dates: First submitted 2017-06-06; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Thrombosis
MeSH Terms: conditions — Thrombosis | interventions — Mutation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warfarin resistant patients (Experimental): Genetic Mutations
  Interventions: Diagnostic Test: Genetic Mutations
- Control (Placebo Comparator): Genetic Mutations
  Interventions: Diagnostic Test: Genetic Mutations

INTERVENTIONS:
Diagnostic Test: Genetic Mutations — By next generation sequencing

SUMMARY:
As drug response is a complex trait in the majority of cases using an optimal starting dose for an individual may reduce the time taken to reach a stable INR, and reduce the risk of having either a high INR (with a risk of bleeding) or a low INR (with a risk of thrombosis)

DETAILED DESCRIPTION:
The results of this project will benefit in (1) Identification of novel features or mutation types in warfarin resistance genomes. (2) To determine whether other polymorphisms in noncoding regions or their unique haplotype combinations contribute to the variability in the maintenance dose of warfarin, and (3)personalization of the drug and deciding the correct dose from the start.

ELIGIBILITY:
Inclusion Criteria:

* Patients with thrombosis and warfarin resistance

Exclusion Criteria:

* less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-06-06 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
number of patients with genetic polymorphism | 6 months
  patients with abnormal polymorphisms

CONTACTS AND LOCATIONS:
Overall Officials: Amr Gawaly, Consultant, Principal Investigator — Hematology Dept. - Tanta University; Said Hammad Abdou, Prof, Principal Investigator — Clinical Pathology dept.- Tanta University; Enas Abdul-Raouf, Lecturer, Study Director — Biology and Genetics- Tanta University; Abdelaziz Zidane, Lecturer, Study Chair — Genetics-Damanhour University
Locations (1):
- Sherief Abd-Elsalam, Cairo, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided